CLINICAL TRIAL: NCT00157066
Title: Effects of Vitamin D Supplementation on Antimycobacterial Immunity: A Randomised Trial
Brief Title: Effects of Vitamin D Supplementation on Antimycobacterial Immunity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Barts & The London NHS Trust (Other)
Collaborators: Imperial College London (Other); University of Cape Town (Other); Newham Chest Clinic, London E7 8QP, UK (Unknown); Northwick Park Hospital, Harrow, UK (Other); Department of Clinical Biochemistry, Homerton Hospital, London E9 6SR, UK (Other); Environmental Health Department, London Borough of Newham, London E15 4SF, UK (Unknown); Wellcome Trust (Other)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: AM1
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2007-01-08 (Estimated); Status verified 2007-01

CONDITIONS: Tuberculosis
Keywords: Latent tuberculosis infection; Active tuberculosis infection
MeSH Terms: conditions — Tuberculosis; Latent Tuberculosis | interventions — Ergocalciferols

INTERVENTIONS:
Drug: Ergocalciferol

SUMMARY:
The purpose of this study is to determine how vitamin D supplementation (ergocalciferol) affects the immune response to mycobacterial infection.

ELIGIBILITY:
Inclusion Criteria:

* Adult
* Tuberculosis (TB) contact or TB patient

Exclusion Criteria:

* Pregnancy
* Breastfeeding
* Hyperparathyroidism
* Sarcoidosis
* Renal failure
* HIV infection

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 230
Dates: Start 2002-12; Study Completion 2006-09

PRIMARY OUTCOMES:
Bacillus Calmette-Guerin (BCG) lux whole blood assay

SECONDARY OUTCOMES:
Antigen-stimulated whole blood interferon gamma production

CONTACTS AND LOCATIONS:
Overall Officials: Adrian R Martineau, B Med Sci, MBBS, DTM&H, MRCP, Principal Investigator — Centre for Health Sciences, Barts and The London, QMUL
Locations (1):
- Tuberculosis Clinic, Newham Chest Clinic, London, United Kingdom

REFERENCES:
- [Derived] Martineau AR, Wilkinson RJ, Wilkinson KA, Newton SM, Kampmann B, Hall BM, Packe GE, Davidson RN, Eldridge SM, Maunsell ZJ, Rainbow SJ, Berry JL, Griffiths CJ. A single dose of vitamin D enhances immunity to mycobacteria. Am J Respir Crit Care Med. 2007 Jul 15;176(2):208-13. doi: 10.1164/rccm.200701-007OC. Epub 2007 Apr 26. PMID 17463418